CLINICAL TRIAL: NCT02383940
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of LX4211 in Young Adult Patients With Type 1 Diabetes Mellitus and Elevated Hemoglobin A1C
Brief Title: Efficacy and Safety of Sotagliflozin in Young Adult Patients With Type 1 Diabetes Mellitus and Elevated Hemoglobin A1C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LX4211.1-204-T1DM; LX4211.204 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2015-02-19; First posted 2015-03-10 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Two placebo-matching sotagliflozin tablets, once daily, orally, before the first meal of the day for 12 weeks.
  Interventions: Drug: Placebo
- Sotagliflozin 400 mg (Experimental): Sotagliflozin 400 milligram (mg) (two 200 mg tablets), once daily, orally, before the first meal of the day for 12 weeks.
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Sotagliflozin — Sotagliflozin 400 mg, once daily before the first meal of the day
  Other Names: LX4211
  Arms: Sotagliflozin 400 mg
Drug: Placebo — Placebo, once daily before the first meal of the day
  Arms: Placebo

SUMMARY:
This Phase 2 study was intended to demonstrate superiority of sotagliflozin versus placebo on Hemoglobin A1C (A1C) reduction at Week 12 in young adult participants with type 1 diabetes mellitus (T1DM) who have poor glycemic control on their current insulin regimen.

ELIGIBILITY:
Inclusion Criteria:

* Participant had given written informed consent.
* Young adult participants >=18 to <=30 years old at Screening, with a confirmed diagnosis of T1DM made at least 1 year prior to informed consent.
* Participants were being treated with insulin or insulin analogue delivered via continuous subcutaneous insulin infusion (CSII) or multiple daily injections (MDI).
* At Screening, must had A1C >= 9.0%.
* Must be willing and able to perform self-monitored blood glucose (SMBG) and complete the study diary.
* Females of childbearing potential must use an adequate method of contraception and had a negative pregnancy test.

Exclusion Criteria:

* Any prior use of LX4211/sotagliflozin.
* Use of antidiabetic agent other than insulin or insulin analogue at the time of screening.
* Use of sodium-glucose cotransporter (SGLT) inhibitors within 8 weeks prior to start of the placebo Run-in Period.
* Chronic systemic corticosteroid use.
* Type 2 diabetes, or severely uncontrolled diabetes mellitus as determined by the Investigator.
* History of diabetic ketoacidosis (DKA) or nonketotic hyperosmolar state within 6 months prior to the Screening Visit.
* History of severe hypoglycemic event within 1 month prior to the Screening Visit.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Sawhney, M.D., Study Director — Lexicon Pharmaceuticals, Inc.
Locations (15):
- United States (15):
  - Lexicon Investigational Site, Tustin, California
  - Lexicon Investigational Site, Aurora, Colorado
  - Lexicon Investigational Site, New Haven, Connecticut
  - Lexicon Investigational Site, Tampa, Florida
  - Lexicon Investigational Site, West Palm Beach, Florida
  - Lexicon Investigational Site, Atlanta, Georgia
  - Lexicon Investigational Site, Roswell, Georgia
  - Lexicon Investigational Site, Indianapolis, Indiana
  - Lexicon Investigational Site, New Orleans, Louisiana
  - Lexicon Investigational Site, Auburn, Maine
  - Lexicon Investigational Site, Boston, Massachusetts
  - Lexicon Investigational Site, Buffalo, New York
  - Lexicon Investigational Site, Wilmington, North Carolina
  - Lexicon Investigational Site, Austin, Texas
  - Lexicon Investigational Site, Salt Lake City, Utah

REFERENCES:
- [Derived] Bode BW, Cengiz E, Wadwa RP, Banks P, Danne T, Kushner JA, McGuire DK, Peters AL, Strumph P, Sawhney S. Effects of Sotagliflozin Combined with Intensive Insulin Therapy in Young Adults with Poorly Controlled Type 1 Diabetes: The JDRF Sotagliflozin Study. Diabetes Technol Ther. 2021 Jan;23(1):59-69. doi: 10.1089/dia.2020.0079. PMID 32640846

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 15 sites in United States between 20 April 2015 and 23 September 2016.
Pre-assignment Details: 147 participants were screened and 87 participants with Type 1 diabetes mellitus who had inadequate glycemic control with insulin therapy alone, were randomized equally into two treatment groups: sotagliflozin 400 milligrams (mg) or placebo.
Groups:
- Sotagliflozin 400 mg: Sotagliflozin 400 mg (two 200 mg tablets), once daily, orally, before the first meal of the day for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 400 mg
Started | 44 | 43
Treated | 42 | 43
Completed | 35 | 40
Not Completed | 9 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Randomized but not treated | 2 | 0
Not completed — Other than specified above | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on modified intent-to treat (mITT) population which included all randomly assigned participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 400 mg | Total
Number analyzed (Participants) | 42 | 43 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.7 (3.55) | 22.8 (4.01) | 22.3 (3.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 19 | 21 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 34 | 41 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Body weight [Mean (Standard Deviation); unit: kilogram (kg)] | 77.27 (14.570) | 83.74 (20.439) | 80.54 (17.975)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] | 26.73 (4.993) | 29.39 (7.214) | 28.07 (6.324)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 11.9 (5.38) | 11.9 (6.16) | 11.9 (5.75)
Insulin Delivery Method [Count of Participants; unit: Participants]
  Continuous Subcutaneous Insulin Infusion (CSII) | 23 | 23 | 46
  Multiple Daily Injections (MDI) | 19 | 20 | 39
Hemoglobin A1C Level in Participants [Count of Participants; unit: Participants]
  <=10 percent (%) | 19 | 18 | 37
  >10 % | 23 | 25 | 48
Baseline daily total insulin [Mean (Standard Deviation); unit: International units per kilogram (IU/kg)] | 0.87 (0.315) | 0.84 (0.264) | 0.86 (0.289)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 12
Description: Baseline was defined as the last value collected prior to the first dose of double-blind study medication. Change was calculated by subtracting baseline value from Week 12 value. Least Square (LS) mean changes from baseline were obtained from mixed model repeated measures (MMRM) model with treatment, randomization strata of insulin delivery (MDI, CSII) and Week-4 A1C (<=10%, >10%), time (study week), and a treatment-by-time interaction as fixed categorical effects, and baseline A1C-by-time interaction as a covariate.
Time Frame: Baseline, Week 12
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of A1C
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 34 | 40
percentage of A1C | -0.99 (0.149) | -1.33 (0.143)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; Between-group comparison was based on MMRM model with treatment, randomization strata of insulin delivery (MDI, CSII) and Week-4 A1C (<=10%, >10%), time (study week), and a treatment-by-time interaction as fixed categorical effects, and baseline A1C-by-time interaction as a covariate; Test type: Superiority; p = 0.10, MMRM — Threshold for significance = 0.05; Least squares mean difference = -0.35, 95% CI 2-sided [-0.76 to 0.06], Standard Error of Mean 0.207 — Difference is sotagliflozin - placebo

2. Secondary Outcome: Change From Baseline in Total Daily Bolus Insulin Dose and Total Daily Basal Insulin Dose at Week 12
Description: The daily bolus and basal insulin doses were calculated as an average of the doses over 3 to 5 days before each visit (Baseline and Week 12). Change was calculated by subtracting baseline value from Week 12 value. LS mean changes from baseline were obtained from MMRM model.
Time Frame: Baseline, Week 12
Population: Analysis included participants from the mITT population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: International Units per day (IU/day)
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 34 | 40
International Units per day (IU/day)
  Total Daily Bolus Insulin Dose | -2.96 (1.945) | -4.89 (1.832)
  Total Daily Basal Insulin Dose | 3.26 (1.262) | 2.03 (1.211)

3. Secondary Outcome: Change From Baseline in 2-hour Postprandial Glucose (PPG) Following a Standardized Mixed Meal at Week 12
Description: A 2-hour PPG sample (plasma) was obtained 2-hours after a standardized Mixed Meal at Baseline (Day 1) and at the visit at Week 12. At Week 12, study drug was to be given within 15 minutes before liquid "Boost®," "Ensure®," or similar nutrition drink product; at baseline, study drug was to be given after the 2-hour post-Mixed Meal PPG sample. Change was calculated by subtracting baseline value from Week 12 value. LS mean changes from baseline were obtained from analysis of covariance (ANCOVA) model.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 32 | 36
milligrams per deciliter (mg/dL) | 0.2 (12.24) | -56.4 (11.61)

4. Secondary Outcome: Change From Baseline in Glycemic Instability by Hyperglycemia (Continuous Glucose Monitoring [CGM] Area Under the Curve [AUC] >150 mg/dL) and Hypoglycemia (CGM AUC <70 mg/dL) Over a 24-hour Period at Week 12
Description: Glycemic instability (mg/dL*minutes/1000) by hyperglycemia/hypoglycemia was measured by CGM AUC outside target range (as a daily average over the week prior to the visit [Baseline and Week 12]) over 24 hours, where outside target range was defined as CGM glucose AUC >150 mg/dL (hyperglycemia) and CGM glucose AUC <70 mg/dL (hypoglycemia). Change was calculated by subtracting baseline value from Week 12 value. LS mean changes from baseline were obtained from MMRM model.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL*minutes/1000
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 28 | 27
mg/dL*minutes/1000
  Glycemic Instability by Hyperglycemia | -5.035 (7.9092) | -27.338 (8.0100)
  Glycemic Instability by Hypoglycemia | 0.221 (0.2508) | 0.428 (0.2528)

5. Secondary Outcome: Change From Baseline in Number of Hypoglycemic Events/Day (<=70 mg/dL) by Self-Monitored Blood Glucose (SMBG) at Week 12
Description: Hypoglycemic event by SMBG was defined as an event in which the fingerstick measurement was <=70 mg/dL. The number of hypoglycemic events per day was calculated as a daily average number of episodes over the week prior to visit (Baseline and Week 12). Change was calculated by subtracting baseline value from Week 12 value. LS mean changes from baseline were obtained from MMRM model.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: events/day
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 35 | 40
events/day | -0.042 (0.0408) | -0.001 (0.0379)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from Baseline (Day 1) until the end of study (up to Week 12).
Description: Analysis was performed on Safety Population defined as all randomly assigned participants who have taken at least 1 dose of study drug.
Arm/Group | Placebo | Sotagliflozin 400 mg
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/43
Serious Adverse Events (participants affected / at risk) | 3/42 | 2/43
Other Adverse Events (participants affected / at risk) | 16/42 | 21/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | Sotagliflozin 400 mg (N=43)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | Sotagliflozin 400 mg (N=43)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Blood ketone body increased (Investigations) | 3 (3) | 8 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (4) | 5 (6)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.